CLINICAL TRIAL: NCT04075877
Title: FOCUS: Feasibility, Acceptability, and Pilot of an Intervention to Improve Functioning in Adolescents With Sickle Cell Disease and Cancer
Brief Title: FOCUS for Pediatric Sickle Cell Disease and Cancer
Acronym: FOCUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Georgia State University (Other)
Responsible Party: Principal Investigator, Laura Mckee, Associate Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FOCUS
Record Dates: First submitted 2019-07-09; First posted 2019-09-03 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-01

CONDITIONS: Pediatric Cancer; Sickle Cell Disease; Quality of Life; Depressive Symptoms; Coping Skills
Keywords: Pediatric cancer; Pediatric Sickle Cell Disease; Quality of Life; Randomized Controlled Trial; Intervention; Photography; Narrative Psychology; Adolescence
MeSH Terms: conditions — Neoplasms; Anemia, Sickle Cell; Depression

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The care provider and the outcomes assessor will be blind to participants' study assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOCUS (Experimental): Participants will complete a baseline survey battery and learn about The Hero's Journey. Starting at hospital discharge for 10 days, they will do the following: 1) identify which stage of The Hero's Journey they are experiencing; 2) take a picture of something good and write a caption describing the picture and provide advice; and 3) take a picture of something difficult or challenging during the day and write a caption for the photo and provide advice.
  Daily text messages will remind participants to take the photographs, write the advice captions, upload both to the server, as well as to take a very brief daily survey. At the conclusion of day 10, participants will be asked to review their photos and captions and provide final advice in the form of a letter to other adolescents with SCD or cancer. Finally, they will complete a post-intervention battery.
  Interventions: Behavioral: FOCUS
- Control (No Intervention): In a 30-min visit (in person or virtual) with adolescents during hospitalizations, we will have participants complete a baseline survey battery.
  Daily text messages will remind participants to take a very brief daily survey. At the conclusion of day 10, participants will complete a post-intervention battery.

INTERVENTIONS:
Behavioral: FOCUS — See prior section.
  Arms: FOCUS

SUMMARY:
Aim. Pilot FOCUS. A pilot randomized controlled trial will compare FOCUS to standard care. Investigators will randomize a total of 60 12- to 18-year-old patients to either FOCUS intervention (n=15 with SCD; n=15 with cancer) or treatment as usual (n=15 with SCD; n=15 with cancer). Randomization will be stratified to match patients based on age, sex, and medical condition (SCD type, cancer type). FOCUS participants will engage in the intervention and complete measures for 10 days post hospital discharge. Control participants will complete similar measures but not receive the intervention. Mixed qualitative and quantitative measures of feasibility, acceptability, and preliminary outcomes will be conducted to evaluate both the intervention and study procedures.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) and cancer are medical conditions in youth that are associated with psychosocial problems including anxiety and depressive symptoms and impaired health-related quality of life. Both SCD and cancer can require a number of treatments and hospitalizations, which negatively impact family relationships, peer functioning, and other life domains. In addition, both conditions and treatments can involve a range of symptoms or side effects (e.g., pain, fatigue, nausea) that interfere with daily life. In other words, patients with SCD and cancer are responsible for gradually learning to manage and live with challenges associated with their medical condition. As such, recent efforts focus on providing psychological interventions to support self-management as an adjunct to standard medical care.

Children and adolescents with SCD and cancer may have limited access to skilled psychologists or may not be able to attend frequent in-person intervention visits to acquire skills to support psychosocial functioning. A critical barrier to helping adolescents with SCD and cancer is that there are few portable interventions that provide assistance outside of the hospital environment.

The goal of this proposal is to pilot test FOCUS (Framing Opportunities and Challenges Using Stories), an innovative and portable intervention designed to improve the psychosocial functioning of adolescents with medical conditions. The intervention involves taking and captioning purposeful photographs that align with The Hero's Journey, a guiding narrative template that chronicles a hero's passage through life's adventures and challenges, culminating in individual strength and transformation (Campbell, 1968). Preliminary data evaluating components of FOCUS revealed significant improvements in mood among healthy adolescents and young adults. Data suggest that reflecting on positive and negative daily events (e.g., via a photograph) and writing about the experiences have profound positive effects on a range of outcomes (e.g., grit, gratitude, functioning). In addition, the investigators intend to share the participants' photographs, stories, and advice on a website for other adolescents with SCD or cancer. Data indicate that prosocial behavior (e.g., providing advice to peers) and social connectedness have a number of positive outcomes. The central prediction is that FOCUS will be acceptable and feasible to deliver and that pilot data will reveal improvements in participants' psychosocial health. Achieving these aims will provide the foundational data needed for federal grant applications to evaluate FOCUS with a larger pediatric sample and other patient populations, powered to identify outcomes and mechanisms of change.

Aim. Pilot FOCUS. A pilot randomized controlled trial will compare FOCUS to standard care. Investigators will randomize a total of 60 12- to 18-year-old patients to either FOCUS intervention (n=15 with SCD; n=15 with cancer) or treatment as usual (n=15 with SCD; n=15 with cancer). Randomization will be stratified to match patients based on age, sex, and medical condition (SCD type, cancer type). FOCUS participants will engage in the intervention and complete measures for 10 days post hospital discharge. Control participants will complete similar measures but not receive the intervention. Mixed qualitative and quantitative measures of feasibility, acceptability, and preliminary outcomes will be conducted to evaluate both the intervention and study procedures.

ELIGIBILITY:
Inclusion Criteria:

* 1) diagnosis of sickle cell disease, any hemoglobin type or diagnosis of leukemia, lymphoma, or solid tumor
* 2) inpatient at CHOA
* 3) 12-18 years of age
* 4) English speaking
* 5) owns a smartphone with camera.

Exclusion Criteria:

* 1) report of active psychosis or active suicidal ideation in the adolescents
* 2) significant documented developmental delay, autism spectrum disorder, or significant intellectual impairment, as these comorbidities may confound the study aims by impacting the dependent measures.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Life Satisfaction | Change from baseline to post-intervention at 10 days
  PROMIS (Patient-Reported Outcomes Measurement Information System) Pediatric Item Bank v1.0 - Life Satisfaction - Short Form 8a; Forrest, C. B., Devine, J., Bevans, K. B., Becker, B. D., Carle, A. C., Teneralli, R. E., … Ravens-Sieberer, U. (2018). Development and psychometric evaluation of the PROMIS Pediatric Life Satisfaction item banks, child-report, and parent-proxy editions. Quality of life research : an international journal of quality of life aspects of treatment, care and rehabilitation, 27(1), 217-234. doi:10.1007/s11136-017-1681-7; Scores range from 8-40, with higher scores representing more life satisfaction
Depression | Change from baseline to post-intervention at 10 days
  PROMIS (Patient-Reported Outcomes Measurement Information System) Pediatric Item Bank v2.0 - Depressive Symptoms - Short Form 8a; Irwin, D. E., Stucky, B., Langer, M. M., Thissen, D., Dewitt, E. M., Lai, J. S., … DeWalt, D. A. (2010). An item response analysis of the pediatric PROMIS anxiety and depressive symptoms scales. Quality of life research : an international journal of quality of life aspects of treatment, care and rehabilitation, 19(4), 595-607. doi:10.1007/s11136-010-9619-3; Scores range from 8-40, with higher scores representing more depression
Anxiety | Change from baseline to post-intervention at 10 days
  PROMIS (Patient-Reported Outcomes Measurement Information System) Pediatric Item Bank v2.0 - Anxiety Symptoms - Short Form 8a; Irwin, D. E., Stucky, B., Langer, M. M., Thissen, D., Dewitt, E. M., Lai, J. S., … DeWalt, D. A. (2010). An item response analysis of the pediatric PROMIS anxiety and depressive symptoms scales. Quality of life research : an international journal of quality of life aspects of treatment, care and rehabilitation, 19(4), 595-607. doi:10.1007/s11136-010-9619-3; Scores range from 8-40, with higher scores representing more anxiety
Meaning and Purpose | Change from baseline to post-intervention at 10 days
  PROMIS (Patient-Reported Outcomes Measurement Information System) Pediatric Item Bank v2.0 - Meaning and Purpose - Short Form 8a; Christopher B Forrest, Katherine B Bevans, Ania Filus, Janine Devine, Brandon D Becker, Adam C Carle, Rachel E Teneralli, JeanHee Moon, Ulrike Ravens-Sieberer, Assessing Children's Eudaimonic Well-Being: The PROMIS Pediatric Meaning and Purpose Item Banks, Journal of Pediatric Psychology, jsz046, https://doi.org/10.1093/jpepsy/jsz046; Scores range from 8-40, with higher scores representing more meaning and purpose
Positive Affect | Change from baseline to post-intervention at 10 days
  PROMIS (Patient-Reported Outcomes Measurement Information System) Pediatric Item Bank v2.0 - Positive Affect - Short Form 8a; Forrest, C. B., Ravens-Sieberer, U., Devine, J., Becker, B. D., Teneralli, R., Moon, J., … Bevans, K. B. (2018). Development and Evaluation of the PROMIS® Pediatric Positive Affect Item Bank, Child-Report and Parent-Proxy Editions. Journal of happiness studies, 19(3), 699-718. doi:10.1007/s10902-016-9843-9; Scores range from 8-40, with higher scores representing more positive affect
Functional Disability | Change from baseline to post-intervention at 10 days
  Functional Disability Inventory (FDI)
Mindfulness | Change from baseline to post-intervention at 10 days
  Child and Adolescence Mindfulness Measure (CAMM)
Approach to Dealing with Adversity | Change from baseline to post-intervention at 10 days
  Shift and Persist Measure

SECONDARY OUTCOMES:
Resilience | Change from baseline to post-intervention at 10 days
  Conner-Davidson Resilience Scale - 10; Davidson, J. R. T. & Connor, K. M. Connor-Davidson Resilience Scale (CD-RISC) Manual. Unpublished. 06-01-2018 and partly accessible at www.cd-risc.com.Total Score Range 0-40, with higher scores reflecting higher resilience
Social Connectedness | Change from baseline to post-intervention at 10 days
  Social Connectedness and Social Assurance Scale; Lee, R. M., & Robbins, S. B. (1995). Measuring belongingness: The social connectedness and the social assurance scales. Journal of Counseling Psychology, 42, 232-241; Using the Social Connectedness Factor only; 8 items; Range 8-48, with higher scores reflecting higher levels of social connectedness and belongingness

OTHER OUTCOMES:
Executive Functioning | Change from baseline to post-intervention at 10 days
  PROMIS Cognitive Function
Prosocial Behavior | Change from baseline to post-intervention at 10 days
  Self-Report of Aggression and Social Behavior Measure, Prosocial Behavior subscale

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey L Cohen, PhD, Principal Investigator — Georgia State University; Laura G McKee, Principal Investigator — Georgia State University
Locations (2):
- United States (2):
  - Georgia State University, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No